CLINICAL TRIAL: NCT06729424
Title: "Living an Active Life with Osteoporosis" - a Digital Patient Education Program on Osteoporosis. a Feasibility/pilot Study As Part of the PATOS Project (Patient Education in Osteoporosis).
Acronym: PilotPATOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Linkoeping University (Other Government); Sormland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Anna Spangeus, Associate Professor, Senior Consultant, University Hospital, Linkoeping
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PilotPATOS
Record Dates: First submitted 2024-12-07; First posted 2024-12-11 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Osteoporosis
Keywords: osteoporosis; patient education; eHealth; self-care
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Digital patient education program (Experimental): Digital patient education program for 5 weeks
  Interventions: Device: Digital patient education program

INTERVENTIONS:
Device: Digital patient education program — The education consists of 8 modules including main themes within osteoporosis, with content aiming to promote behavioural changes including psychoeducation and behavioural activation.

SUMMARY:
In this feasibility and pilot study, the investigators aim to evaluate the effectiveness and safety of a digital patient education program for individuals with osteoporosis. The study involves a 5-week intervention period during which participants will have access to the digital education program. Patients will be assessed both before and after the intervention.

The digital patient education program comprises eight modules covering essential topics related to osteoporosis self-care. The program includes both psychoeducation and support for behavioral changes. Patients will progress through the program at their own pace.

The name of the digital patient education program is: program is: "Att leva ett aktivt liv med benskörhet" (translated to english "Living an Active Life with Osteoporosis")

ELIGIBILITY:
Inclusion Criteria:

* Osteoporosis diagnosis with or without a previous low-energy fracture
* Age > 50 years
* Women and men
* Basic computer skills

Exclusion Criteria:

* Patients with difficulty understanding the Swedish language to the extent that they cannot comprehend the content of the patient education program.
* Cognitive impairment/dementia where the patient is not deemed to understand the implications of study participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (HRQoL) - generic | 6 weeks
  Assessed with RAND-36 (Research and Development questionnaire). The RAND-36 compromises 36 items with two to six response options according to an ordinal scale. Eight health domains are assessed, coded, scored and summarised to derive the domains. The scores are transformed into a 0-100 scale. Zero indicates the worst possible HRQoL and 100 the best.
Health-related quality of life (HRQoL) - generic | 6 weeks
  Assessed with EQ-5D-5L. The EQ5D covers 5 dimensionsand. In addition to these dimensions, the EQ-5D includes a visual analogue scale (VAS) where respondents rate their overall health on a scale.
Self-Care in osteoporosis | 6 weeks
  Assessed with 26 questions in 5 domains (medication, diet, physical training, fall risk, ergonomy). Questions covering knowledge, motivation, opportunities and behaviour.
Patient enablement instrument (PEI) | 6 weeks
  The patient enablement instrument (PEI) is used to measure the patient's perceived change in ability to understand and cope with his or her health issues after the treatment period and contains six items. The text "As a result of the participating in the Osteoporosis School, do you feel that you are …" is followed by six items; 1) able to cope with life, 2) able to understand your illness, 3) able to cope with your illness, 4) able to keep yourself healthy, 5) confident about your health, and 6) able to help yourself. The following five alternative answers were used for each statement; much better/much more, better/more, same, less/worse and not applicable. The PEI point for much better/much more is 2; for better/more is 1; and for same, less/worse or not applicable is 0. These points are added and thus the total PEI score ranges between 0 (worst score) and 12 (best score).
Fear of falling | 6 weeks
  Assessed with Falls Efficacy Scale-International (FES-I). The FES-I is a 16-item questionnaire used to measure the level of concern about falling during social and physical activities inside and outside the home. Each item I scored on a 4-point Likert scale ranging from (1 = not concerned, and 4= very concerned). The item scores are summed up to a total score ranging from minimum 16 to maximum 64 with higher the score higher being the concern for falling.
Fear avoidance beliefs regarding physical activity | 6 weeks
  The Fear-Avoidance Beliefs Questionnaire physical activity subscale (FABQ_FA) include 4 questions about physical activity. Agreement with each statement is rated on a 7-point Likert Scale (0= completely disagree, to 6= completely agree), and a total score is calculated (maximum of 24) with higher scores indicates stronger fear avoidance beliefs.
Illness perception | 6 weeks
  Assessed with the Brief-Illness Perception Questionnaire BIPQ which is an 8-item questionnaire that assesses cognitive and emotional representation of illness. Each item is rated on a 0-10 scale with higher scores indicating a more threatening perception of the illness. The total score is calculated by summing the scores and range between 0-80 with higher scores indicate worse illness perception.
Self-reported physical activity, alcohol consumption and smoking | 6 weeks
  The questionnaire (Hälsobladet) is used in clinical routine in Sweden to assess self-reported lifestyle habits on a weekly basis
Self-reported pain and intake of pain medication | 6 weeks
  Self-reported pain was assessed both regarding intensity (NRS 0-10) and frequency as well as medication intake.
Self-reported fall and balance | 6 weeks
  Self-reported fall during the last year as well as perceived balance was assessed (NRS 0-10)
Maximal walking speed | 6 weeks
  Walking speed was assessed with patients walking 10 meters at a maximal walking speed.
Hand-strength | 6 weeks
  Assessed in sitting position with the Jamar both right and left side.
Chair Sit to stand (30 sec) | 6 weeks
  The maximal number of sit to stand during 30 seconds.
Measure of hyperkyfosis | 6 weeks
  With patients in upright standing distance between C7 and wall, as well as between tragus of the ear to wall was evaluated.
Timed-loading standing test | 6 weeks
  Ability to stand up with weights (1-0.5 kg) in both arms during a maximum of 2 minutes
One-leg standing with eyes opened | 6 weeks
  Assessed for both right and left legs and a maximum of 60 seconds
One-leg standing with eyes closed | 6 weeks
  Assessed for both right and left legs and a maximum of 60 seconds.
Walking on a line | 6 weeks
  Patients were asked to take a maximum of 15 steps forward on a line and then a maximum of 15 steps backwards on a line.
Timed-up and go (TUG) | 6 weeks
  Patients were asked to stand up from sitting and walt 3 meters, turning around, walk back and sit again. Time was measured in seconds.

OTHER OUTCOMES:
Activity Pattern | 6 weeks
  Activity pattern will be measured with activPAL™ in a subset of patients (n=10). The activPAL™ will be used recording physical activities during 7 days (including time spent lying, sitting, standing and stepping).

CONTACTS AND LOCATIONS:
Locations (1):
- Linköping University Hospital, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No